CLINICAL TRIAL: NCT03535103
Title: A Randomized, Open-label, Two-Period, Two-Crossover Study to Compare the Safety and Pharmacokinetics of Recombinant Human Follicle Stimulating Hormone Injection (LM001) and Gonal-F® in Healthy Female Volunteers
Brief Title: Study on the Safety and Pharmacokinetics of LM001 and Gonal-F® in Healthy Women
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alphamab Jilin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KNJR-2018-001
Record Dates: First submitted 2018-05-02; First posted 2018-05-24 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — follitropin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Experimental): Gonal-F®
  Interventions: Drug: Gonal-F®
- ARM B (Experimental): LM001
  Interventions: Drug: LM001

INTERVENTIONS:
Drug: Gonal-F® — A single Subcutaneous injection, 225IU
  Other Names: Follitropin alfa
  Arms: ARM A
Drug: LM001 — A single Subcutaneous injection, 225IU
  Other Names: Follitropin alfa
  Arms: ARM B

SUMMARY:
Brief Summary: LM001 is a recombinant human Follicle Stimulating Hormone (r-hFSH) Injection, which is proposed for Assisted Reproductive Technology (ART). This is a randomized, open-label, two-period, two-crossover study to evaluate the safety and pharmacokinetics of recombinant human follicle stimulating hormone injection (LM001), compared with Gonal-F®, both given subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Agreed to take effective contraceptive measures during and 6 months after the end of the study period.
3. Age between 18 to 40 years (inclusive).
4. Body weight ≥45 kg, body mass index (BMI) of ≥18 and ≤28 kg/m2,
5. Regular menstruation cycle (25 to 34 days, inclusive).
6. Normal findings in sex hormone examinations, including FSH, LH, prolactin (PRL), estradiol (E2), progesterone (P), testosterone (T) unless the investigator considers an abnormality to be clinically irrelevant for this study.

Exclusion Criteria:

1. Smoke ≥5 cigarettes or the equivalent per day within 3 months prior to the study
2. History of hypersensitivity to FSH, or hypersensitivity to luteinizing hormone releasing hormone agonist or something like that.
3. Historic abuse of alcoholic beverages and drugs (Drink 14 units of alcohol/week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine.
4. Taken any liver enzyme activity relative drug within 28 days prior to the screening.
5. Take any prescription drug, OTC drug, vitamin product or herbal medicine within 14 days prior to the screening.
6. Taken special diets (including pitaya, mango, grapefruit, etc.) or have strenuous exercise, or something affect the absorption, distribution, metabolism, excretion, etc. of the drug within 2 weeks prior to the study.
7. Major changes in diet or exercise habits recently
8. Participation in a clinical study within 3 months prior to the study.
9. Acute disease or combination therapy from the screening to the beginning time of the study.
10. Take any alcoholic product within 48 hours prior to the study.
11. Take chocolate, any caffeine-containing or xanthine-rich food or drinks within 48 hours prior to using the drug;
12. Blood donation or massive blood losing (>450mL) within 3 months prior to the screening;
13. Viral hepatitis (including hepatitis B and hepatitis C), HIV, and Treponema pallidum positive.
14. History of significant diseases such as circulatory, endocrine, neurological, reproductive, digestive, and respiratory systems, hematology, immunology, psychiatry, and metabolic abnormalities, or past or current medical history that could interfere with the test results, eg subjects with or have suffered from hypothyroidism, adrenocortical insufficiency and hyperprolactinemia, polycystic ovary syndrome, and ovarian dysfunction, premature ovarian failure (POI) or primary ovarian failure, unexplained uterine bleeding, hypothalamic or pituitary tumors, ovarian, uterine or breast cancer, history of thrombosis, history of malignancy;
15. Baseline of serum FSH ≥15 IU/L.
16. History of ovarian hyperstimulation syndrome (OHSS).
17. Other abnormalities judged by researchers of the study
18. Abnormal physical examination and clinical significance judged by researchers of the study
19. Abnormal vital signs and clinical significance judged by researchers of the study.
20. Abnormal laboratory tests with clinically relevance.
21. Abnormal electrocardiogram [ECG] findings.
22. III/IV class endometriosis, submucous myoma of uterus, endocrine abnormalities within 6 months prior to the study.
23. Abnormal imaging examination and clinical significance judged by researchers of the study, such as with a uterine fibroid diameter ≥ 40 mm.
24. Pregnancy or lactation period.
25. Alcohol screening positive.
26. Urine drug screening positive

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Maxmum observed serum concentration (Cmax) of LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Maxmum observed serum concentration (Cmax) of LM001＆Gonal-f® in healthy Chinese female subjects.
Adjusted geometric means of area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUC(0-T))for LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Adjusted geometric means of area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUC(0-T))for LM001＆Gonal-f® in healthy Chinese female subjects.

OTHER OUTCOMES:
Time of Maxmum observed serum concentration (Tmax) of LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Time of Maxmum observed serum concentration (Tmax) of LM001＆Gonal-f® in healthy Chinese female subjects.
Serum clearance(CL) of of LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Serum clearance(CL) of of LM001＆Gonal-f® in healthy Chinese female subjects.
Adjusted geometric means of area under the serum concentration-time curve from time zero extrapolated to infinite time(AUC(INF))for LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Adjusted geometric means of area under the serum concentration-time curve from time zero extrapolated to infinite time(AUC(INF))for LM001＆Gonal-f® in healthy Chinese female subjects.
Serum Half-life(T-HALF)of LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Serum Half-life(T-HALF)of LM001＆Gonal-f® in healthy Chinese female subjects.
Apparent volume of distribution（VD）)of LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Apparent volume of distribution（VD）)of LM001＆Gonal-f® in healthy Chinese female subjects.
Expression of terminal clearance rate constant（λ z ）of LM001＆Gonal-f® in healthy Chinese female subjects. | within 0.5h pre-dose, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168 hours post-dose.
  Expression of terminal clearance rate constant（λ z ）of LM001＆Gonal-f® in healthy Chinese female subjects.
Number of Participants with Abnormal Labortory Values and/or Adverse Events that are realated to treatment(SAEs) and AEs of special interest. | From screening to up to 16 days.
  Number of Participants with Abnormal Labortory Values and/or Adverse Events that are realated to treatment(SAEs) and AEs of special interest.